CLINICAL TRIAL: NCT04055935
Title: Evaluation of the Effect of Full Thickness Mucoperiosteal Flap Versus Low Level Laser in Orthodontic Tooth Movement Acceleration
Brief Title: Full Thickness Mucoperiosteal Flap Versus Low Level Laser in Orthodontic Tooth Movement Acceleration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohsena Ahmad, Assistant lecturer of orthodontics, Al-Azhar University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: Doctor's degree research
Record Dates: First submitted 2019-07-30; First posted 2019-08-14 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Mesial Movement of Teeth
MeSH Terms: conditions — Mesial Movement of Teeth | interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: split mouth study design, side intervention and other side for control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- full thickness mucoperiosteal flap (Experimental): A full thickness mucoperiosteal flap (FTMPF) was reflected on FTMPF side at the maxillary canine/premolar region by the same surgeon for all patients following the same procedures.
  Interventions: Procedure: elevation of full thickness mucoperiosteal flap
- low level laser therapy (Experimental): LLLT was done using a diode soft laser (Epic X, BioLase, USA). It is a semiconductor diode soft laser. Active medium is In-Ga-As with 940nm wave length
  Interventions: Device: low level laser therapy
- Control for Full thickness mucoperiosteal flap (No Intervention): Control for Full thickness mucoperiosteal flap, in which canine retraction was done in a conventional method
- control for Low level laser therapy group (No Intervention): Control for Low level laser therapy , in which canine retraction was done in a conventional method

INTERVENTIONS:
Procedure: elevation of full thickness mucoperiosteal flap — A free gingival sulcular incision was done from the distal surface of maxillary second premolar to the mesial side of the maxillary canine. A releasing oblique incision was done including the interdental papilla between maxillary canine and lateral incisor extending to the mucogingival junction just beyond the attached mucosa. The flap reflection extended beyond the canine root apex. A FTMPF reflection was done with mucoperiosteal elevator. Free sulcus incision was done to allow elevation of palatal mucosa by tunneling technique on the palatal gingiva of maxillary canine.
  Arms: full thickness mucoperiosteal flap
Device: low level laser therapy — LLLT was done using a diode soft laser (Epic X, BioLase, USA). It is a semiconductor diode soft laser. Active medium is In-Ga-As with 940nm wave length. LLLT protocol was using active laser tip (bleaching tip)
  Arms: low level laser therapy

SUMMARY:
This study aimed to evaluate the effect of using full thickness mucoperiosteal flap (FTMPF) elevation only versus low level laser therapy (LLLT) on acceleration of orthodontic tooth movement.

DETAILED DESCRIPTION:
This study was a split mouth design study included 32 side according to sample size calculation. Those sides were divided into 2 groups. Group 1divided into (group 1a: 8 sides with FTMPF, group 1b:8 sides control). Group 2(group 2 a: 8 sides with LLLT, group 2b: 8 sides control). Extraction of the first maxillary premolars followed by canine retraction in the extraction space with maximum anchorage were indicated. FTMPF was elevated from the mesial interdental papilla of maxillary canine to the mesial interdental papilla of second maxillary premolar. LLLT was applied at 3,7,14,28.56 days of retraction. During retraction study model for all patients were taken at 2ed, 6th, 14th,16th weeks and at the end of retraction (I1,I2,I3,I4,I5 or overall interval). 3D laser scanning and digital superimposition was done to measure the rate of canine retraction and anchorage loss.

ELIGIBILITY:
Inclusion Criteria:

* o Free of any syndromes affecting the head region or any craniofacial injuries.

  * No history of previous orthodontic treatment
  * All of the permanent dentition present excluding third molars.
  * Good oral hygiene before starting treatment.
  * Cases indicated for extraction of the maxillary first premolars and canine retraction into the extraction space with maximum anchorage.
  * Malocclusion cases that allow initial stage of leveling and alignment without extraction.

Exclusion Criteria:

* o Patients with systemic diseases especially bleeding disorders and osteoporosis.

  * History of administration of corticosteroids, exogenous hormones and non-steroidal anti-inflammatory drugs (all drugs interfere with OTM).
  * Presence of previous history of oral surgeries in maxillary arch.

Ages: 15 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
rate of orthodontic tooth movement acceleration determination by measuring the rate of maxillary canine retraction | the rate of retraction( distance from the first day of retraction to the end of retraction/ time)) it was with total time frame 24 weeks for starting of retraction
  measure the rate of canine retraction on series of study models

SECONDARY OUTCOMES:
clinical mesial movement of first maxillary molar measured by millimeter on the 3D model | t0(start of canine retraction) to 24 months
  amount of mesial movement of first maxillary molar after 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Mohsena a arazik, orthodontist, Principal Investigator — Al-Azhar University
Locations (1):
- Faculty of dentistry ,Al-Azhar Univerisity, Cairo, Naser City, Egypt

IPD SHARING:
Plan to Share IPD: Yes
the data will be shared the weekly rate and distance of canine retraction, the amount of maxillary canine mesial movement and the periodontal pocket depth around the maxillary canine
Supporting Information: Study Protocol, SAP, ICF
Time Frame: by today,()30July 2019
Access Criteria: Google drive
URL: https://drive.google.com/open?id=1VGIPJwCULeNnotdILJ4o5znvMF5pdPIw

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/35/NCT04055935/SAP_000.pdf
  • Study Protocol (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/35/NCT04055935/Prot_001.pdf